CLINICAL TRIAL: NCT05011552
Title: Self-Compassion, Health, and Empowerment: A Feasibility Intervention Study for Chinese Immigrant Women With Intimate Partner Violence in the U.S.
Brief Title: Feasibility Study for Abused Chinese Immigrant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Yang Li, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00001645
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Intimate Partner Violence; Depression; Anxiety; PTSD
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental)
  Interventions: Behavioral: Self-Compassion, Health, and Empowerment (SHE)
- The control group (Placebo Comparator)
  Interventions: Behavioral: The Control Condition

INTERVENTIONS:
Behavioral: Self-Compassion, Health, and Empowerment (SHE) — The SHE intervention includes 8 weekly sessions and 24-hour access to the intervener for any additional support needed. The first and last sessions will be delivered over the phone with the woman based on a brochure. The brochure describes the four major components: a) IPV information, b) Danger Assessment, c) Safety Planning, and d) Resources. It will be discussed with the woman in an interactive manner so that the woman is encouraged to describe her experiences and choose her options as they proceed. Session 2-7 focus on providing mental health self-care resources, which are deep breathing, progressive muscle relaxation, visualization, general introduction and overview of self-compassion, mindfulness, and loving-kindness.
  Arms: The intervention group
Behavioral: The Control Condition — Women randomized to the control group will be provided with the same brochure and mental health care resources.
  Arms: The control group

SUMMARY:
Intimate partner violence (IPV) is a serious social and public health issue. In the U.S., more than 1 in 3 women experience physical or sexual violence, and/or stalking by an intimate partner during their lifetime. IPV has significant physical and mental health consequences such as injury, chronic pain, and depression. Chinese immigrants have been overlooked and underserved and represent an especially vulnerable group of IPV victims, as they are less likely to seek help through IPV service agencies, women's shelters, hospitals, or law enforcement. Effective IPV intervention programs that are culturally appropriate, accessible, and acceptable are essential to this underserved population. However, no studies have been conducted with abused Chinese immigrant women to help them deal with IPV and reduce mental health consequences.

Therefore, the study adapted a structured IPV intervention from the Domestic Violence Enhanced Home Visitation Program (DOVE) as well as incorporate self-compassion and relaxation techniques for Chinese immigrant women experiencing IPV. The intervention is called Self-Compassion, Health, and Empowerment (SHE). The study will test the feasibility and acceptability of the SHE to reduce IPV and improve mental health well-being for abused Chinese immigrant women residing in the US.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and female, self-identify as Chinese, reside in the U.S., have been in an intimate relationship at time of participation, and have experienced IPV within the current relationship.

Exclusion Criteria:

* Women are excluded if they report substance use or suicidality or having been in mental health care for severe mental illness.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Intimate Partner Violence | It will be assessed at baseline before the start of the 8-week intervention.
  The Revised Conflict Tactics Scales (CTS2)
Intimate Partner Violence | It will be assessed immediately after the 8-week intervention.
  The Revised Conflict Tactics Scales (CTS2)
Intimate Partner Violence | It will be assessed 2 months after the 8-week intervention.
  The Revised Conflict Tactics Scales (CTS2)
Depression | It will be assessed at baseline before the start of the 8-week intervention.
  The Patient Health Questionnaire-9 (PHQ-9)
Depression | It will be assessed immediately after the 8-week intervention.
  The Patient Health Questionnaire-9 (PHQ-9)
Depression | It will be assessed 2 months after the 8-week intervention.
  The Patient Health Questionnaire-9 (PHQ-9)
Anxiety | It will be assessed at baseline before the start of the 8-week intervention.
  The Generalized Anxiety Disorder-7 (GAD-7)
Anxiety | It will be assessed immediately after the 8-week intervention.
  The Generalized Anxiety Disorder-7 (GAD-7)
Anxiety | It will be assessed 2 months after the 8-week intervention.
  The Generalized Anxiety Disorder-7 (GAD-7)
Posttraumatic Stress Disorder (PTSD) | It will be assessed at baseline before the start of the 8-week intervention.
  The PTSD Checklist for DSM-5 (PCL-5)
Posttraumatic Stress Disorder (PTSD) | It will be assessed immediately after the 8-week intervention.
  The PTSD Checklist for DSM-5 (PCL-5)
Posttraumatic Stress Disorder (PTSD) | It will be assessed 2 months after the 8-week intervention.
  The PTSD Checklist for DSM-5 (PCL-5)

SECONDARY OUTCOMES:
Number of Safety Behaviors Taken by Participants | It will be assessed at baseline before the start of the 8-week intervention.
  The Intimate Partner Violence Strategies Index
Number of Safety Behaviors Taken by Participants | It will be assessed immediately after the 8-week intervention.
  The Intimate Partner Violence Strategies Index
Number of Safety Behaviors Taken by Participants | It will be assessed 2 months after the 8-week intervention.
  The Intimate Partner Violence Strategies Index
Self-Compassion | It will be assessed at baseline before the start of the 8-week intervention.
  The Self-Compassion Scale-Short Form (SCS-SF)
Self-Compassion | It will be assessed immediately after the 8-week intervention.
  The Self-Compassion Scale-Short Form (SCS-SF)
Self-Compassion | It will be assessed 2 months after the 8-week intervention.
  The Self-Compassion Scale-Short Form (SCS-SF)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas At Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li Y, Rhee H, Bullock LFC, McCaw B, Bloom T. Self-Compassion, Health, and Empowerment: A Pilot Randomized Controlled Trial for Chinese Immigrant Women Experiencing Intimate Partner Violence. J Interpers Violence. 2024 Apr;39(7-8):1571-1595. doi: 10.1177/08862605231207624. Epub 2023 Oct 30. PMID 37902465